CLINICAL TRIAL: NCT07301684
Title: Analysis of a Multimodal Physiotherapy Treatment in Pediatric and Adolescent Cancer Survivors: A Randomized Clinical Trial
Brief Title: Physiotherapy in Pediatric Oncology
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: University of Seville, Spain (Unknown)
Responsible Party: Principal Investigator, Miriam Linero Bocanegra, Physiotherapy, University of Seville
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2025-11-24; First posted 2025-12-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: pediatrics; oncology
MeSH Terms: conditions — Neoplasms | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: Three intervention arms:
  1. Therapeutic physical exercise
  2. Therapeutic physical exercise + electrotherapy
  3. Therapeutic physical exercise + gamified game
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP EXERCISE (Active Comparator)
  Interventions: Other: Therapeutic physical exercise
- GROUP ELECTROTHERAPY (Active Comparator)
  Interventions: Other: Therapeutic physical exercise + electrotherapy
- GROUP EXERGAMING (Active Comparator)
  Interventions: Other: Therapeutic physical exercise + gamified game

INTERVENTIONS:
Other: Therapeutic physical exercise — Specific therapeutic exercise intervention based on FITT parameters and working with aerobic, anaerobic, and breathing exercises.
  Arms: GROUP EXERCISE
Other: Therapeutic physical exercise + electrotherapy — Specific therapeutic exercise intervention based on FITT parameters and working with aerobic, anaerobic, and breathing exercises. Combined with the application of electrical waves for neurostimulation of the quadriceps muscles.
  Arms: GROUP ELECTROTHERAPY
Other: Therapeutic physical exercise + gamified game — Specific therapeutic exercise intervention based on FITT parameters and focusing on aerobic, anaerobic, and breathing exercises. Combined with the application of gamified exercise to improve treatment adherence in these young populations.
  Arms: GROUP EXERGAMING

SUMMARY:
The objective of this clinical trial is to determine whether therapeutic physical exercise combined with electrotherapy and exercise gaming improves rehabilitation outcomes in pediatric and adolescent cancer patients.

The main questions it aims to answer are:

Does the combination of therapeutic physical exercise plus muscle strengthening and therapeutic physical exercise plus gamification, compared to a single exercise intervention, improve patient condition? Does gamified exercise improve treatment adherence? Does electrotherapy improve muscle activity when used in muscle strengthening mode? Researchers will test the application of the described modalities and assess improvements in variables such as cardiorespiratory fitness, physical activity self-efficacy, pain, balance, joint range of motion, physical activity level, cancer-related fatigue, quality of life, anxiety-depression, sleep, kinesophobia, and social status.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed cancer treatment and are currently in remission, referred by their oncologist.
* Children and adolescents aged 3 to 16 years.
* Patients with a stable medical condition, without severe or acute complications related to cancer or its treatments.
* Patients whose informed consent (from parents/legal guardians, in this case, as they are minors) has been obtained to participate in this study.
* Patients with sufficient physical capacity to tolerate the activities proposed by the program.

Exclusion Criteria:

* Severe comorbidities: neuromuscular, cardiovascular, or respiratory diseases that prevent participation in the exercise program or interfere with the assessment of physical function.
* Incompatible medical treatments: patients currently receiving active treatments or with medical contraindications for electrotherapy or participation in exercise programs.
* Severe psychological issues: children with severe psychological disorders or cognitive disabilities that may hinder understanding and participation in the sessions.
* Visual impairments: patients with visual problems will not be able to participate, as this may interfere with the analysis of results related to the use of devices and video games for exercise.
* Participation in other clinical trials: patients already involved in other research that could interfere with the results of this study.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Strength | 6 month
  30-second sit-to-stand test to measure lower extremity muscle performance: is a functional measure of lower-limb strength in which an individual stands up and sits down from a chair as many times as possible within 30 seconds. If the test is reported using a numerical score, it corresponds to the total number of completed sit-to-stand repetitions, where the minimum value is 0, the maximum value depends on the person's performance, and higher scores indicate better lower-body strength and functional capacity.
Cardiorespiratory function | 6 month
  6-minute walk test: is a widely used assessment of cardiorespiratory function in which an individual is instructed to walk as far as possible along a flat, measured course for six minutes. When reported numerically, the score corresponds to the total distance walked in meters, with a minimum value of 0 meters, no fixed maximum (as it depends on individual performance), and higher distances indicating better cardiorespiratory capacity and endurance.
Physical activity self-efficacy | 6 month
  The five-item Physical Activity Self-Efficacy Scale (PASE): is a brief self-report measure that evaluates an individual's confidence in their ability to engage in physical activity under various challenging circumstances. Scores are obtained by summing responses to the five items, each typically rated on a scale from 1 (low confidence) to 5 (high confidence), yielding a minimum total score of 5 and a maximum of 25. Higher scores indicate better self-efficacy for maintaining physical activity.
Pain level | 6 month
  Visual Analog Scale (VAS): is a simple, widely used measure for assessing the intensity of subjective experiences such as pain, fatigue, or discomfort. It typically consists of a 10-centimeter horizontal line anchored by verbal descriptors at each end-for example, 0 = "no pain" and 10 = "worst imaginable pain." The respondent marks a point on the line that represents their perceived intensity. The minimum score is 0, the maximum score is 10, and higher scores indicate a worse symptom intensity.
Balance | 6 month
  Pediatric Berg Balance Scale (BBS): is a performance-based assessment designed to measure functional balance in children through 14 tasks such as standing, turning, and reaching. Each item is scored from 0 (inability to perform) to 4 (independent, best performance), producing a minimum total score of 0 and a maximum of 56. Higher scores indicate better balance ability and greater functional stability.
Ankle dorsiflexion ROM | 6 month
  Goniometer: is an instrument used to measure the range of motion (ROM) of a joint. For ankle dorsiflexion, the goniometer is positioned with the axis at the lateral malleolus, the stationary arm aligned with the fibula, and the movable arm along the fifth metatarsal. Measurements are reported in degrees, with a typical minimum of 0° and a maximum depending on the individual, usually around 20° for dorsiflexion. Higher values indicate greater ankle dorsiflexion ROM, reflecting better joint flexibility.
Weight | 6 month
  Tanita DC-439 MA
Height | 6 month
  Harpender stadiometer
BMI | 6 month
  weight/height 2
Bone mineral density | 6 month
  Ultrasound (QUS Model: Bone Mineral Densiometer, (OSTEOSYS, BETTER PRODUCTS FOR BETTER LIFE, n.d.))
Muscle circumferences (upper arm, waist, hip, and thigh) | 6 month
  Tape measure

SECONDARY OUTCOMES:
Physical activity levels | 6 month
  Accelerometry Test: is an objective method for assessing physical activity levels by having an individual wear an accelerometer device, usually on the wrist, hip, or ankle, which records movement intensity and duration. Data are typically reported as average counts per minute, steps per day, or minutes spent in different activity intensities (e.g., sedentary, light, moderate, vigorous). Minimum values can be 0, and the maximum depends on the individual's activity level. Higher values indicate greater levels of physical activity.
Cancer-related fatigue | 6 month
  PedsQL™ Multidimensional Fatigue Scale: is a self-report questionnaire designed to assess fatigue in children across three domains: General Fatigue, Sleep/Rest Fatigue, and Cognitive Fatigue. Items are scored on a 5-point Likert scale (0 = "Never" to 4 = "Almost Always"), which are then reverse-scored and transformed to a 0-100 scale, with higher scores indicating less fatigue and better functioning. The minimum total score is 0, the maximum is 100, and higher scores reflect lower fatigue levels.
Cancer-related Quality of life | 6 month
  PedsQL™ Pediatric Quality of Life Questionnaire (Spanish version for Children and Adolescents with Heart Disease (PedsQL™)): is a self-report instrument that assesses health-related quality of life across multiple domains, including physical, emotional, social, and school functioning. Items are rated on a 5-point Likert scale (0 = "Never" to 4 = "Almost Always"), which are then reverse-scored and transformed to a 0-100 scale. The minimum total score is 0, the maximum is 100, and higher scores indicate better health-related quality of life.
Anxiety-depressive symptoms | 6 month
  The Children's Depression Inventory (CDI): is a self-report questionnaire designed to assess depressive symptoms in children and adolescents aged 8 to 18 years. It consists of multiple items scored on a 0-2 scale, with the minimum total score of 0 and a maximum total score of 54. Higher scores indicate more severe depressive symptoms.
  Childhood Anxiety Sensitivity Index (CASI): is a self-report measure that evaluates the fear of anxiety-related sensations in children. Items are rated on a 3-point scale (1 = "None" to 3 = "A lot"), with a minimum total score of 18 and a maximum of 54. Higher scores reflect greater anxiety sensitivity.
Sleep | 6 month
  Pediatric Sleep Questionnaire (PSQ): is a parent- or caregiver-reported tool used to screen for sleep-related problems in children, including sleep-disordered breathing, snoring, and daytime sleepiness. Items are typically scored as "Yes" = 1, "No" = 0, or "Don't know" = missing. The total score is calculated as the proportion of positive responses, with a minimum of 0 and a maximum of 1. Higher scores indicate more sleep-related problems.
Kinesiophobia | 6 month
  Kinesiophobia Questionnaire for Children (KQC) adapted from the Tampa Scale for Kinesiophobia (TSK): is a self-report instrument designed to assess fear of movement or reinjury in children. Items are typically scored on a 4-point Likert scale (1 = "Strongly Disagree" to 4 = "Strongly Agree"), with a minimum total score of 13 and a maximum of 52. Higher scores indicate greater kinesiophobia, reflecting a stronger fear of movement or activity due to pain or injury.
Treatment Adherence | 6 month
  Exercise Adherence Rating Scale: is a self-report questionnaire used to assess an individual's adherence to prescribed exercise programs. Items are typically scored on a 5-point Likert scale (0 = "Completely Disagree" to 4 = "Completely Agree"), with a minimum total score of 0 and a maximum of 24 for the adherence section. Higher scores indicate better adherence to the exercise regimen.
Social Support | 6 month
  Social Support Questionnaire for Children (SSQ-C): is a self-report instrument designed to assess the perceived availability and satisfaction with social support in children. It includes items asking about the number of supportive people (availability) and satisfaction with support. Scores are typically summarized as average number of supporters per item and average satisfaction rating, with minimum values of 0 and maximum values depending on the scale used for satisfaction (often 6 or 7). Higher scores indicate greater perceived social support and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: MANOLO M ALBORNOZ CABELLO, FISIOTERAPEUTA, Principal Investigator — FACULTAD DE ENFERMERÓIA, FISIOTERAPIA Y PODOLOGÍA
Locations (1):
- Facultad de Enfermería, Fisioterapia y Podología, Seville, Spain

IPD SHARING:
Plan to Share IPD: No